CLINICAL TRIAL: NCT03248323
Title: A Prospective Study: the Value of Using Parametric Color Coding of Digital Subtraction Angiography and Flat-panel Detector Computed Tomography Parenchymal Blood Volume Imaging in the Endovascular Treatment of Infrapopliteal Arterial Occlusive Diseases
Brief Title: A Prospective Study: the Value of Using iFlow and PBV in the Endovascular Treatment of Infrapopliteal Arterial Occlusive Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A03968
Record Dates: First submitted 2017-05-09; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2016-06

CONDITIONS: Arterial Occlusive Diseases
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (1):
- pre-con
  Interventions: Radiation: dyna-pbv

INTERVENTIONS:
Radiation: dyna-pbv

SUMMARY:
Color coded blood flow and blood perfusion techniques are applied to the endovascular treatment of infrapopliteal arterial occlusion,to establish a method of quantitative evaluation of blood flow and tissue perfusion,to improve the level of calculation of condition and curative effect. So as to establish a new complete evaluation system of infrapopliteal arterial occlusive disease, to guide clinical further. At the same time establish a digital information platform for clinical, lay the foundation for the large research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are diagnosed as lower limb atherosclerosis occlusion from June 2016 to June 2018 in our centre;
2. All participating patients provided written informed consent and willing to participate;
3. aged 40 years and more;
4. the class of lower ischemia is upon 4;
5. below-the-knee arteries stenosis or occlusion is indicated by duplex or computed tomographic angiography;
6. there is no heavy stenosis in superficial femoral artery (stenosis<30%), or short length lesion(length≤5cm, stenosis≥30%);
7. infection or ulceration don't happen in the area of surgery;
8. below the inguinal ligament arteries don't have the history of bypass or interventional surgery.

Exclusion Criteria:

1. disagree and refuse to the free therapy;
2. lesion length of superior artery is more than 5cm;
3. history of heart dysfunction: congestive heart failure,, myocardial infarction, severe arrhythmia;
4. With severe metabolic disease, renal impairment(serum creatinine>1.4mg/dL, glomerular filtration rate<60) affect the excretion of contrast agents;
5. have the diseases or agents which will reduce the viable of data;
6. allergy to iodinated contrast medium.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These new technologies are performed in the treatment of patients older than 40 years. They present with rest pain, intermittent claudication, ulceration or gangrenous. Some of them have the risk factors of CLI, as hypertension, diabetes, hyperlipidemia or smoking. They are referred to our vascular service for CLI-infrapopliteal artery occlusion. Computed tomographic angiography discloses the occlusive lesion in anteriortibial, posterior tibial or peroneal arteries.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
patency rate | 1 year
  We compare the change of blood flow velocity and blood perfusion volume before and after the recanalization of infrapopliteal arteries to assess the initial patency rate. While we test the ankle brachial index and toe brachial index at 3 , 6, 12 months, lower extremity arterial ultrasound at 6 mouths and computed tomographic angiography in 1 year to evaluate the patency of one year.

SECONDARY OUTCOMES:
wound healing rate | 1 year
  This is to evaluate the prognosis of patients who with the foot ulcer.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Shao J, Ma J, Lai Z, Yu X, Li K, Xu L, Chen J, Wang C, Cao W, Liu X, Yuan J, Liu B. Impaired pedal arch affects the treatment effect in patients with single tibial artery revascularization demonstrated by intraoperative perfusion. Quant Imaging Med Surg. 2022 Jun;12(6):3204-3212. doi: 10.21037/qims-21-801. PMID 35655837